CLINICAL TRIAL: NCT05023941
Title: Optimization Strategy for the Prevention of Acute Mountain Sickness by Remote Ischemic Preconditioning Combined With Acetazolamide
Brief Title: Optimization Strategy for the Prevention of AMS by RIPC Combined With Acetazolamide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ji Xunming,MD,PhD (Other)
Responsible Party: Sponsor-Investigator, Ji Xunming,MD,PhD, VP, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: RIPC-Acet-AMS
Record Dates: First submitted 2021-08-15; First posted 2021-08-27 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Acute Mountain Sickness
Keywords: Acute Mountain Sickness; Acetazolamide; Remote Ischemic Preconditioning
MeSH Terms: conditions — Altitude Sickness | interventions — Acetazolamide

STUDY DESIGN:
Masking Description: Due to the nature of the procedure, it was not possible to blind subjects to the intervention of medicine or RIPC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Medicine Group (Active Comparator): Start orally take Acetazolamide 2 days before entering the hypoxic room.
  Interventions: Drug: Acetazolamide
- RIPC Group (Active Comparator): Start RIPC training twice daily, 6 days before entering the hypoxic room.
  Interventions: Device: Doctormate® (twice daily for 6 days)
- Rapid RIPC Group (Experimental): Start RIPC training forth daily, 3 days before entering the hypoxic room.
  Interventions: Device: Doctormate® (forth daily for 3 days)
- Combined Group (Experimental): Medicine + Rapid RIPC
  Interventions: Drug: Acetazolamide; Device: Doctormate® (forth daily for 3 days)
- Control Group (No Intervention): Subjects do not receive specific interventions before entering the hypoxic room.

INTERVENTIONS:
Drug: Acetazolamide — Start orally take acetazolamide 125mg twice daily, 2 days before entering the hypoxic chamber. Subjects will enter the hypoxic room at 9am on the third day. At that time, the subject should have taken the drug 5 times.
  Arms: Combined Group; Medicine Group
Device: Doctormate® (twice daily for 6 days) — Start RIPC training twice daily, 6 days before entering the hypoxic chamber. RIPC will be induced by Renqiao Remote Ischemic Conditioning Device (Doctormate®). Each training will be comprised of 5 cycles of bilateral upper limb ischemia and reperfusion, which will be induced by 2 cuffs placed around the upper arms respectively and inflated to 200mmHg for 5 minutes followed by 5 minutes of reperfusion by cuff deflation. Subjects will enter the hypoxic room at 9am on the seventh day. At that time, the subject should have finished 13 times of RIPC training.
  Arms: RIPC Group
Device: Doctormate® (forth daily for 3 days) — Start RIPC training forth daily, 3 days before entering the hypoxic chamber. RIPC will be induced by Renqiao Remote Ischemic Conditioning Device (Doctormate®). Each training will be comprised of 5 cycles of bilateral upper limb ischemia and reperfusion, which will be induced by 2 cuffs placed around the upper arms respectively and inflated to 200mmHg for 5 minutes followed by 5 minutes of reperfusion by cuff deflation. Subjects will enter the hypoxic room at 9am on the forth day. At that time, the subject should have finished 13 times of RIPC training.
  Arms: Combined Group; Rapid RIPC Group

SUMMARY:
The primary objective of the study will be to determine whether rapid remote limb ischemic preconditioning (RIPC) combined with acetazolamide can further reduce the incidence of acute mountain sickness (AMS) during the 6-hour hypoxic chamber.

DETAILED DESCRIPTION:
The current measures to prevent acute mountain sickness (AMS) mainly include drug prevention and non-drug prevention. Acetazolamide is a drug approved by the U.S. FDA for the prevention and treatment of AMS. Remote limb ischemic preconditioning (RIPC) can also reduce the incidence of AMS as a non-durg method, with a strategy of 2 times/day training for 1 week reducing the incidence of AMS in 6 hours from 40% to 30%. The objective of this study is to determine whether rapid RIPC training combined with acetazolamide can further reduce the incidence of AMS. In this study, subjects will be divided into 5 groups: medicine group (acetazolamid 125mg bid, 2 days before entering the hypoxic room), RIPC group (RIPC training twice daily, 6 days before entering the hypoxic room), rapid RIPC group (RIPC training forth daily, 3 days before entering the hypoxic room), combined group (rapid RIPC training plus acetazolamide) and controlled group. RIPC training, completed by Renqiao Remote Ischemic Conditioning Device (Doctormate®), will be comprised of 5 cycles of bilateral upper limb ischemia and reperfusion, which will be induced by 2 cuffs placed around the upper arms respectively and inflated to 200mmHg for 5 minutes followed by 5 minutes of reperfusion by cuff deflation. After the intervention, subjects will be exposed to 4500m altitude in a normobaric hypoxic chamber for 6 hours. The incidence of AMS and other data will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* People who live in plain areas all year round and have not been to an altitude of 1500 meters or more in the past 30 days;
* Sign the informed consent form voluntarily.

Exclusion Criteria:

* Chronic physical or mental diseases, including hypertension, diabetes, coronary heart disease, cerebrovascular disease, chronic obstructive pulmonary disease, migraine, anxiety, depression, insomnia, etc.;
* The female is pregnant or in the period of preparing for pregnancy or breast-feeding;
* Have a history of smoking;
* Have a history of thrombosis in the upper limbs;
* Severe damage to local soft tissues of upper limbs, fractures, etc.;
* Allergic to sulfa;
* Are taking one or more drugs;
* Past laboratory tests suggest hypokalemia, hyponatremia, or liver and kidney damage;
* Patients unsuitable for enrollment in the clinical trial according to investigators decision making.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 252 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
The incidence of acute mountain sickness. | 6 hours after entering the hypoxic room.
  The diagnosis of acute mountain sickness is based on '2018 Lake Louise Acute Mountain Sickness Score' , 'Acute Mountain Sickness-Cerebral Scores',etc. All subjects should finish the questionnaires to evaluate the total incidence.
The severity of acute mountain sickness. | 6 hours after entering the hypoxic room.
  The diagnosis of acute mountain sickness is based on '2018 Lake Louise Acute Mountain Sickness Score' , 'Acute Mountain Sickness-Cerebral Scores',etc. All subjects should finish the questionnaires to evaluate the total incidence.
Fingre pulse oximetry of the subjects. | 6 hours after entering the hypoxic room.
  Fingre pulse oximetry using pocket pulse oximeters will be noted.

SECONDARY OUTCOMES:
Blood pressure of the subjects. | 6 hours after entering the hypoxic room.
  Including systolic and diastolic pressure.
Heart rate of the subjects. | 6 hours after entering the hypoxic room.
Respiratory rate of the subjects. | 6 hours after entering the hypoxic room.

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, MD.PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu M, Jiao X, Li R, Li J, Wang L, Wang L, Wang Y, Lv C, Huang D, Wei R, Wang L, Ji X, Guo X. Effects of acetazolamide combined with remote ischemic preconditioning on risk of acute mountain sickness: a randomized clinical trial. BMC Med. 2024 Jan 2;22(1):4. doi: 10.1186/s12916-023-03209-7. PMID 38166913